CLINICAL TRIAL: NCT07278141
Title: Study Protocol: Effects of Combined Resistance Training and Dual-Task Interventions on Physical, Oculomotor, and Executive Functions in Older Adults With Mild Cognitive Impairment. A Randomized Controlled Trial
Brief Title: Effects of Resistance and Dual-Task Training on Physical, Oculomotor, and Executive Functions in Older Adults With MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas, Chile (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Ivonne Andrea Jorquera Cáceres, Physical therapist, MSc, Universidad Santo Tomas, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4126162
Record Dates: First submitted 2025-05-08; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Physical Function; Executive Function (Cognition); Saccadic Eye Movements
Keywords: combination training; Dual-Task; Physical-Cognitive Training; aging; older adult; Timed Up & Go; executive function; Resistance Training

STUDY DESIGN:
Intervention Model Description: The intervention period will last 8 weeks, with therapeutic intervention programs consisting of 3 weekly sessions. The older adults (OA) of EGR group will receive a minimum of 20 sessions, with a maximum of up to 24 sessions.
  Each resistance training session will last one hour and will consist of three parts: Preparation (joint mobility and basic movements for warm-up), Resistance Training (Implementing added weight exercises), Cool Down (breathing exercises and stretches). Weight exercises will focus on the flexor/extensor groups of the elbow and the flexor/extensor groups of the knee, through bilateral leg presses, unilateral knee extensions, and bilateral elbow flexo-extensions. These exercises will be performed in 3 sets of 8 repetitions for each trained muscle group.
  The combined resistance training group with dual-task exercises (EGRD) will follow the same exercise protocol and additionally incorporate memory and arithmetic tasks. The CG will receive the usual care.
Who Masked: Outcomes Assessor
Masking Description: Due to the study design, proper blinding is not feasible, as it is a non-pharmacological within-subject design. The intervention is visible to both the participants and the investigators administering it. To mitigate this issue, in accordance with the CONSORT extension for non-pharmacological trials (Boutron et al., 2017), the study's hypothesis is concealed from the participants, and the outcomes assessor at the beginning and the end of the intervention will be blinded to the participants' intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group EGR (Experimental group resistance exercises) (Experimental): EGR will receive only anaerobic therapeutic exercises (resistance exercises) for 8 weeks, with 3 sessions per week. The exercises will focus on the elbow flexor/extensor groups and the knee flexor/extensor groups, using a bilateral leg press, unilateral knee extensions, and bilateral elbow flexion-extension exercises, performed in 3 sets of 8 repetitions for each trained muscle group.
  Interventions: Procedure: Anaerobic therapeutic exercises (resistance exercise)
- The EGRD group (Experimental group: resistance exercise plus dual tasks) (Experimental): The EGRD group (experimental group: resistance exercise plus dual tasks) will receive 8 weeks of anaerobic therapeutic exercises (resistance exercises) combined with dual tasks during sessions. They will perform the same exercise protocol as the EGR group and concurrently add memory and arithmetic tasks during the exercises.
  Interventions: Combination Product: Anaerobic therapeutic exercises (resistance exercise) plus Dual Task
- The CG Group (control group) (No Intervention): The control group (CG) will receive usual health care during the intervention period; however, they will receive the best evaluated therapeutic intervention at the end of the study.

INTERVENTIONS:
Procedure: Anaerobic therapeutic exercises (resistance exercise) — The intervention period will last 8 weeks, with 3 sessions per week. Each resistance training session will last one hour and will consist of three parts: the first part will include joint mobility and basic preparatory movements; the second part will involve the resistance training itself (with added weight); and finally, the third part will feature breathing exercises and stretches as a cool-down. Weighted exercises will focus on the elbow flexor/extensor groups and the knee flexor/extensor groups through bilateral leg presses, unilateral knee extensions, and bilateral elbow flexion-extension exercises, performed in 3 sets of 8 repetitions for each muscle group trained. The training intensity for the first two weeks will be set at 60% of 1RM and will then be increased to the target intensity (80% of 1RM) by at least week 7 of the training. To ensure that the training program is progressive, a 1RM strength evaluation will be performed every two weeks, to adjust the training load.
  Arms: Intervention Group EGR (Experimental group resistance exercises)
Combination Product: Anaerobic therapeutic exercises (resistance exercise) plus Dual Task — The anaerobic (resistance) exercise training group combined with dual tasks will follow the same protocol as the previously described anaerobic therapeutic exercise training and will additionally incorporate memory and arithmetic tasks concurrently during the exercises. The intervention period will also last 8 weeks, with 3 sessions per week, and each training session will last one hour (Pantoja-Cardoso et al. 2023).
  Arms: The EGRD group (Experimental group: resistance exercise plus dual tasks)

SUMMARY:
The goal of this clinical trial is to determine the effect of a combined therapeutic intervention program with anaerobic exercises (resistance exercises) and dual tasks on the physical, oculomotor, and executive functions of older adults with mild cognitive impairment.

The main questions it aims to answer are:

• How effective will a therapeutic intervention program combining resistance exercises with dual tasks be in improving the physical, oculomotor, and executive functions of older adults with mild cognitive impairment living in the community? Researchers will compare the effectiveness of a resistance exercise training program combined with dual tasks versus a resistance-only exercise training program to see if it improves the physical, oculomotor, and executive functions of older adults with mild cognitive impairment

Participants Will:

* Receive resistance exercises, resistance exercises combined with dual tasks. or the standard health care. The intervention programs will consist of 3 weekly sessions over 8 weeks.
* Before the start and after the completion of the programs, they will be evaluated using a battery of tests. This includes sociodemographic and general health background, physical fitness tests, as well as assessments of executive functions and oculomotor Saccadic movements and anti-saccadic error.
* be required to sign a consent form.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted with two experimental groups and one control group. The target population will be older adults with mild cognitive impairment living in the communities of Arica (Chile) and Valencia (Spain). All participants must score between 10 and 25 points on the Montreal Cognitive Assessment (MoCA).

The sample size was calculated using statistical software, based on mean differences reported in prior studies on training and dual tasks in older adults. A minimum of 11 participants per group was established, adjusted for a 20% dropout rate, a significance level of 0.01, and a statistical power of 0.9.

In each city, 33 participants (men and women in a 1:1 ratio) will be recruited. Random distribution by gender will assign participants to three groups:

EGR: Resistance exercises only.

EGRD: Resistance exercises combined with dual tasks (cognitive tasks).

CG: Control group, receiving standard health care during the study and, upon completion, the best-evaluated therapeutic intervention.

Procedure The study will last 12 weeks: two weeks for baseline measurements (pre-test), eight weeks for training protocols, and two weeks for final measurements (post-test). Evaluations will include sociodemographic and health data, functional physical condition tests, executive function assessments, and saccadic and anti-saccadic eye movement measures.

Interventions will be conducted at the physiotherapy faculties of the participating universities, supervised by experienced professionals blinded to group allocation. Participants will be asked not to engage in physical exercise outside the study protocols during evaluation weeks.

Hypotheses

Primary: The combined intervention of resistance exercises and dual tasks is more effective than isolated resistance training in improving physical, executive, and oculomotor functions in older adults with mild cognitive impairment.

Secondary: The combined intervention produces greater improvements in executive function tasks (Stroop Test, Corsi Block-Tapping Test, Trail Making Test) compared to resistance training alone.

Intervention Program

The intervention will last eight weeks, with three weekly sessions (20-24 sessions total). Each resistance training session will last one hour, divided into:

Warm-up: Joint mobility and basic movements; Resistance training: Exercises with external load; Cool-down: Breathing exercises and stretching.

Exercises will target flexor and extensor groups of the elbow and knee, including bilateral leg press, unilateral knee extensions, and bilateral elbow flexion/extension. Three sets of eight repetitions will be performed for each muscle group. Training intensity will begin at 60% of one-repetition maximum (1RM) and progress to 80% by week 7, adjusted every two weeks based on new strength evaluations and perceived exertion.

The combined group (EGRD) will follow the same physical protocol, incorporating memory and arithmetic tasks during exercise execution.

Assessment Instruments

Functional physical condition: Timed Up and Go Test (TUG), Short Physical Performance Battery (SPPB), and grip strength measured with a hydraulic dynamometer.

Executive functions: Inhibitory control: Stroop Test, with three conditions (word, color, word-color); Working memory: Corsi Block-Tapping Test (CBTT), assessing visuo-spatial memory sequences; Cognitive flexibility: Trail Making Test (TMT-A and TMT-B), evaluating speed, attention, and alternation.

Oculomotor function: Electrooculography (EOG) will record saccadic and anti-saccadic movements using surface electrodes and controlled visual stimuli.

Statistical Analysis Population data will be presented as means for continuous variables and prevalence for categorical variables, with 95% confidence intervals. Inferential analyses will consider normality and homoscedasticity to determine parametric or non-parametric tests. A blinded researcher will conduct all analyses using IBM SPSS version 27.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 years or older
* Score between 10 and 25 points on the Montreal Cognitive Assessment (MoCA) scale
* Provide informed consent

Exclusion Criteria:

* Visual or auditory disability that impedes communication
* Previous diagnosis of dementia
* Wheelchair use
* Epilepsy
* Progressive or terminal illness
* Depression
* History of alcoholism
* Musculoskeletal or cardiovascular contraindications for strength exercises
* Color blindness
* Dyslexia
* Severe mental or cognitive problems supported by medical reports

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Physical-functional condition - Risk of falls | Baseline, and immediately post-intervention (week 11),
  The physical-functional condition, specifically the risk of falls of participants will be assessed using the Timed Up and Go Test (TUG). Description: Time in seconds required to stand up from a chair, walk three meters, turn, return, and sit down. Unit of Measure: Seconds (s)
Executive function - Inhibitory control | Baseline, and immediately post-intervention (week 11-12)
  Participants' inhibitory control will be assessed using the Stroop Colour Test. Performance will be evaluated through response time. Unit of Measure: Milliseconds (ms)
Oculomotor Function- Saccadic and anti-saccadic oculomotor movement | Baseline, and immediately post-intervention (week 11)
  Saccadic and anti-saccadic eye movements will be assessed using a non-invasive electrooculography (EOG) system (ADInstruments PTK15 EOG model and AD Instruments Brazil PowerLab T26-3079). Two surface electrodes will be placed at the outer canthi of the right and left eyes, with a ground electrode positioned on the forehead. Synchronization between target illumination and EOG signals will be controlled using LabChart software (version 7, Research Ltd.). Performance will be evaluated based on movement latency during visual tasks: left-to-right for saccadic movements and right-to-left for anti-saccadic movements. Unit of Measure: Milliseconds (ms).
Physical - functional condition - Physical function | Baseline, and immediately post-intervention (week 11)
  The Physical-functional condition, specifically Participants' physical function will be assessed with the Short Physical Performance Battery (SPPB).
  Description: Composite score evaluating balance, gait speed, and lower limb strength. Unit of Measure: Points on a scale (0-12).
Physical - functional condition - Grip Strength | Baseline, and immediately post-intervention (week 11)
  The Physical-functional condition, specifically the grip strenght of particiants will be assesment with the JAMAR dynamometer. Description: Maximum grip strength measured with a hydraulic dynamometer. Unit of Measure: Kilograms (kg)
Executive Function - Working Memory | Baseline, and immediately post-intervention (week 11-12)
  Working memory will be assessed using the Corsi Block-Tapping Test (CBTT), administered in both forward and backward conditions. Performance will be evaluated based on response time for each condition. Unit of Measure: Milliseconds (ms)
Executive Function - Cognitive Flexibility | Baseline, and immediately post-intervention (week 11-12)
  Cognitive flexibility will be assessed using the Trail Making Test (TMT). Performance will be evaluated through completion time for Part A (numbers only) and Part B (numbers and letters alternating). Unit of Measure: Miliseconds (ms).

SECONDARY OUTCOMES:
Sociodemographic variable - Age | Baseline
  Age of participants recorded during the first meeting. Unit of Measure: Years
Sociodemographic variable - Sex | Baseline
  Sex of participants recorded during the first meeting. Unit of Measure: Male/Female (categorical variable).
Sociodemographic variables-Educational Level | Baseline
  Highest educational level attained by participants. Unit of Measure: Categorical variable (e.g., primary, secondary, higher education).
Health indicators- Comorbidities | Baseline
  Presence of comorbidities such as hypertension, diabetes, or hypercholesterolemia, collected through validated questionnaires. Unit of Measure: Presence/absence (binary categorical variable).
Anthropometric variable- Body Mass Index (BMI) | Baseline
  BMI calculated according to WHO protocols as weight (kg) divided by height squared (m²). Unit of Measure: kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Jorquera-Caceres I Ivonne, MSc, Study Director — Universidad Santo Tomas, Chile
Locations (2):
- Arica- Chile y Valencia -España, Arica, Arica y Parinacota Region, Chile
- Valencia-Spain, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Personal information and data for all experiments are handled by the personal information manager director of Valencia University. Access to information requires a key that is securely kept and has limited access. These internal checks and balances ensure the security of all data and personal information. After the experimental period ends, the data will be consolidated. Any information linking data backto the participant will be discarded to ensure that the data are truly anonymous.

REFERENCES:
- [Background] Voos MC, Custodio EB, Malaquias J Jr. Relationship of executive function and educational status with functional balance in older adults. J Geriatr Phys Ther. 2011 Jan-Mar;34(1):11-8. doi: 10.1097/JPT.0b013e3181ff2452. PMID 21937887
- [Background] Vandierendonck A. Working memory benchmarks-A missed opportunity: Comment on Oberauer et al. (2018). Psychol Bull. 2018 Sep;144(9):963-971. doi: 10.1037/bul0000159. PMID 30148381
- [Background] Heath M, Weiler J, Gregory MA, Gill DP, Petrella RJ. A Six-Month Cognitive-Motor and Aerobic Exercise Program Improves Executive Function in Persons with an Objective Cognitive Impairment: A Pilot Investigation Using the Antisaccade Task. J Alzheimers Dis. 2016 Oct 4;54(3):923-931. doi: 10.3233/JAD-160288. PMID 27567829
- [Background] Glisky EL, Alexander GE, Hou M, Kawa K, Woolverton CB, Zigman EK, Nguyen LA, Haws K, Figueredo AJ, Ryan L. Differences between young and older adults in unity and diversity of executive functions. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2021 Nov;28(6):829-854. doi: 10.1080/13825585.2020.1830936. Epub 2020 Oct 8. PMID 33028159
- See also: CONSORT 2025 explanation and elaboration: updated guideline for reporting randomised trials — https://www.bmj.com/lookup/doi/10.1136/bmj-2024-081124
- Available data/document: Study Protocol: Study Protocol ACTIVAM — https://alumnossantotomas-my.sharepoint.com/:b:/g/personal/ivonnejorquera_santotomas_cl/EeBXjIa_2FBMivQW63r3zkQBXK4j0X4-TiOdpAqmw_w2sg?e=Fh6PcR — The study protocol is accessible to anyone with the link
- Available data/document: Data Monitoring Committee Charter: Ethics Committee Approval — https://alumnossantotomas-my.sharepoint.com/:b:/g/personal/ivonnejorquera_santotomas_cl/EfT4D7DeqWJKg0G9BoL0JEIBgmCcMobhIPrQMe2MeCZu0g?e=QlrDDK — The file is publicly available via link
- Available data/document: Informed Consent Form: INFORMED CONSENT — https://alumnossantotomas-my.sharepoint.com/:b:/g/personal/ivonnejorquera_santotomas_cl/ETTRNyC4tIpKgXo3bKwcG-EBWanx328fkqIPiudt0LoMvA?e=m8mMB6